CLINICAL TRIAL: NCT04792697
Title: Center for Adolescent Reward, Rhythms and Sleep Project 2
Brief Title: Experimental Manipulation of Sleep and Circadian Rhythms and the Role Played on Reward Function in Teens
Acronym: CARRS-P2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brant Hasler, Associate Professor of Psychiatry, Psychology and Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20030271; 1P50DA046346-01A1 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-04

CONDITIONS: Delayed Sleep Phase Syndrome
Keywords: adolescence; sleep; substance use; reward sensitivity and motivation; circadian phase and alignment; inhibition
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Substance-Related Disorders; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: This study combines Laboratory, Experimental & Longitudinal protocols with 2 initial groups (Early Sleep Timing & Late Sleep Timing). Both groups complete an initial laboratory protocol (baseline). The Late Sleep participants are also randomized to one of two arms (Manipulation or Control) in the experimental protocol (intervention). Early Sleep group does not complete the experimental protocol. Finally, all participants receive follow-up assessments through the life of the grant in the Longitudinal protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance/Extend Manipulation (Experimental): For ~2 weeks, Manipulation participants will advance bedtime and regularize wake time. The first night of the manipulation will be conducted in the lab under tightly-controlled experimental conditions. Participants will then go home and for the next 12 days and will be instructed to:
  * Sleep scheduling-- advance bedtime by 1.5 hours ( + sleep duration)
  * Decrease evening blue light exposure via blue blocker goggles (2 hrs before bed)
  * Increase morning bright light exposure via bright light goggles (30 min after rise)
  * Monitor sleep, mood, and substance use via smartphone-based platform and wrist actigraph
  Interventions: Other: Increase morning bright light; Other: Decrease evening blue light; Behavioral: Sleep Scheduling; Behavioral: Monitor sleep, mood, and substance use
- Control (Active Comparator): Control participants will complete the baseline laboratory study, then maintain their habitual sleep schedules over the next 12 days at home, with no instruction on sleep timing or light exposure. Control participants will complete smartphone-and text-based assessments and wear an actigraphy watch to monitor their sleep, behavior and sleep habits thereby controlling for effort.
  Interventions: Behavioral: Monitor sleep, mood, and substance use

INTERVENTIONS:
Other: Increase morning bright light — Participants will wear Re-Timer bright glasses for 30 minutes each morning upon rising
  Arms: Advance/Extend Manipulation
Other: Decrease evening blue light — Participants will wear tinted glasses that block blue wavelength light for 2 hours before bed
  Arms: Advance/Extend Manipulation
Behavioral: Sleep Scheduling — Participants will advance their bedtime by 1.5 hours and regularize their wake time
  Arms: Advance/Extend Manipulation
Behavioral: Monitor sleep, mood, and substance use — Participants will complete smartphone-based sleep, mood, and substance use monitoring

SUMMARY:
Adolescence is a time of heightened reward sensitivity and greater impulsivity. On top of this, many teenagers experience chronic sleep deprivation and misalignment of their circadian rhythms due to biological shifts in their sleep/wake patterns paired with early school start times. Many studies find that this increases the risk for substance use (SU). However, what impact circadian rhythm and sleep disruption either together or independently have on the neuronal circuitry that controls reward and cognition, or if there are interventions that might help to modify these disruptions is unknown. Project 2 (P2) of the CARRS center will test an innovative and mechanistic model of brain circuitry that uses multi-method approaches, takes a developmental perspective, and incorporates key sleep and reward constructs.

DETAILED DESCRIPTION:
Substance use (SU) and substance use disorders (SUD) pose devastating health, financial, and societal costs. The incidence of SU and SUDs increases across adolescence, making this sensitive developmental period one of both heightened risk-and heightened opportunity for prevention and intervention. However, to develop effective interventions investigators need to identify novel and modifiable risk factors and mechanisms for SUD. Sleep and circadian rhythm disturbances are such risk factors, and the reward system, with its increasing sensitivity during adolescence, provides a plausible mechanistic substrate. The focus on sleep, circadian rhythms, and reward system function is particularly salient given the extensive, parallel development of these systems during adolescence, and the plausible linkages between sleep and circadian rhythms, reward function, and SUD risk.

Late sleep timing, short sleep duration and circadian misalignment are associated with increased substance use in teenagers and young adults. The central hypothesis of the Center for Adolescent Reward, Rhythms and Sleep (CARRS) is that adolescent development acts on underlying sleep and circadian traits to modify homeostatic sleep drive, circadian phase, and circadian alignment, which in turn impact cortico-limbic functions critical to SU risk (e.g., reward and cognitive control). Investigators further hypothesize that specific manipulations of sleep and circadian rhythms during adolescence will affect reward responsivity and cognitive control in either positive or negative directions. These manipulations will provide experimental support for our model, and proof of concept for novel clinical interventions to reduce the risk of SU and SUDs.

Most previous studies have examined individual components of circadian rhythms, sleep, and reward function in adolescence. Project 2 (P2) of CARRS will test an innovative and mechanistic model of brain circuitry that uses multi-method approaches, takes a developmental perspective, and incorporates key sleep and reward constructs. Most notably, P2 improves upon past observational work by testing an experimental intervention that manipulates sleep and circadian rhythms to directly examine its impact on reward function and cognitive control.

P2 will study 150 adolescents (age 13-15, 50% female) across two key sleep phenotypes: early sleep timing (low risk, n=50) and late sleep timing (high risk, n=100). All participants will complete the observational study: 2 weeks of home sleep monitoring (actigraphy & sleep diary), followed by an overnight laboratory visit to assess self-report, behavioral, and neuroimaging (fMRI) tasks tapping cognitive control and reward function, as well as circadian phase via salivary melatonin and molecular rhythms via hair follicles. The Late group will continue to the experimental study, each participant randomized to manipulation or attentional control conditions (n=50 each). Investigators will probe whether advancing sleep/circadian timing and extending sleep duration via sleep scheduling and chronotherapeutic approaches (reducing PM light exposure; administering AM bright light) improves sleep, circadian, and neurobehavioral function relevant to SUD risk. Finally, repeated 6-month follow-up assessments of sleep and SU for all participants are included to examine longitudinal associations.

ELIGIBILITY:
Inclusion Criteria:

* Typically enrolled in a traditional high-school with synchronous learning (in-person or online synchronous learning, but not cyber- or home-schooling) [school closures during the COVID-19 pandemic are an exception to this]
* Physically and psychiatrically healthy
* Provision of written informed consent and assent
* Additional inclusion criterion for Experimental protocol: Meets operational definition of late sleep timing (>10:50PM habitual bedtime)

Exclusion Criteria:

* History of alcohol, cannabis, or illicit drug use in the past month, or greater than monthly use in the past year
* Significant or unstable acute or chronic medical conditions
* Frequent headaches or migraines
* History of seizures
* Current serious psychiatric disorder (e.g., depressive disorder, bipolar disorder, eating disorder, psychotic disorder diagnosis, alcohol use disorder or substance use disorder) that would interfere with completion of study procedures
* Current syndromal sleep disorders other than insomnia and delayed sleep phase disorder
* MRI contraindications (i.e., absence of metal in the body, claustrophobia)
* Medications that increase sensitivity to blue light/photosensitizing medications, including psychiatric neuroleptic drugs, psoralen drugs, antiarrhythmic drugs, etc.
* Changes to psychotropic medication regimen in the 2 weeks prior to enrollment, and/or major changes to medications during the study protocol
* If participants have an average bedtime that is later than 3:00AM or an average wake time later than 11:00AM they may be excluded from the study
* Participants should be EXCLUDED for other sleep disorders that require ongoing treatment
* Participants should be EXCLUDED for other sleep disorders that cause significant distress or impairment, per DSM 5 criteria in the Sleep SCID.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weekday Sleep Duration--Actigraphy & Diaries | Baseline (2 Weeks), T2 (2 weeks)
  Total Sleep Time as determined by wrist actigraphy data & sleep diaries (averaged across weekdays during 2 weeks at T1 and 2 weeks at T2)
Circadian Timing-Dim Light Melatonin Onset | Baseline Overnight Visit (T1) & T2 Overnight Visit(2 weeks later). Always on a Friday.
  Circadian Timing as determined by dim light melatonin onset during saliva sampling using the 4pg/ml threshold.
Circadian Alignment | Baseline overnight (T1), T2 overnight (2 weeks after T1)
  Circadian alignment is operationalized as the interval between the dim light melatonin onset (DLMO) and sleep midpoint based on the prior two nights of actigraphy data.
Reward motivation (Behavioral) | Baseline overnight (T1) vs. T2 overnight (2 weeks after T1)
  Assessed by adjusted average pumps on Balloon Analogue Risk Task, a computerized measure of risk taking behavior in which participants are presented with a series of balloons and offered the chance to earn money by pumping each balloon up by clicking a button. The adjusted average only includes non-burst trials.
Behavioral Inhibition | Baseline overnight (T1) vs. T2 overnight (2 weeks after T1). Always on a Friday.
  Accuracy on Cued Go/No-Go Task, specifically correct response (withholding response) on No-Go trials following an incongruent Go cue
Neural correlates of Impulse control | Baseline overnight (T1) vs. T2 overnight (2 weeks after T1). Always on a Friday.
  Activation within the Executive Control Network during the Stop Signal Task, a computerized an fMRI behavioral task. Specifically, activation is defined as bold signal in regions of the Executive Control Network on unsuccessful Stop trials versus successful Go trials. Higher values represent increased activity to unsuccessful Stop versus successful Go trials.
Neural correlates of Reward Anticipation | Baseline overnight (T1) vs. T2 overnight (2 weeks after T1). Always on a Friday.
  Activation within the reward network during the Monetary Incentive Delay task, a computerized an fMRI behavioral task. Specifially, activation is defined as bold signal in regions of the reward network (from NeuroSynth), on reward anticipation trials (large reward) versus neutral (no money) trials. Higher values represent increased reactivity to reward, as compared to neutral trials.
Neural Correlates of Reward Receipt | Overnight visits at end of T1 & T2 (two weeks after T1)
  Monetary Incentive Delay Task: Win Outcome vs No Win contrast within the reward network (from Neurosynth). Higher values represent increased reactivity to reward wins, as compared to neutral trials.

SECONDARY OUTCOMES:
Cannabis use | Continuously every 6 months for up to 5 years
  Days of cannabis use on Timeline Follow Back interview administered during the baseline interview and in self-report surveys every 6 months.
Alcohol Use | Continuously every 6 months for up to 5 years
  Days of alcohol use on Timeline Follow Back interview administered during baseline interview and every six months via self-report

CONTACTS AND LOCATIONS:
Overall Officials: Brant Hasler, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Current and future investigators, both internal and external, may have access to de-identified data; however only group data would be shared.